CLINICAL TRIAL: NCT05437133
Title: Reliability and Validity of Self-reported Adherence to Elbow Orthosis Wearing Time Using Concealed Temperature Sensors
Brief Title: Reliability and Validity of Self-reported Adherence to Elbow Orthosis Wearing Time
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 12567
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Elbow Injury; Elbow Fracture; Elbow Arthritis
MeSH Terms: conditions — Elbow Injuries; Elbow Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Custom fabricated elbow extension orthosis — custom low temperature thermoplastic orthosis (Splint) holding the elbow in maximum extension at night

SUMMARY:
The purpose of this study is to validate whether the use of a self-reported diary for orthosis use is accurate and valid. We will insert a temperature gauge into the orthosis during fabrication that measures temperature to an accuracy of one degree Celcius. This sensor is about the size of a watch battery, and patients will be told that it is measuring the force of stretch applied to the elbow, while in fact, it is measuring the amount of time that the orthosis is being worn. The temperature of the skin while wearing the orthosis heats up the sensor, and we can accurately predict (within 5 minutes of accuracy) how long the orthosis is worn each day.

We will have patients also fill out a self-report diary outlining how long they are wearing the orthosis each day, and compare these times to the measurements taken by the sensor. As secondary outcomes, we will look at whether the orthoses improve elbow range of motion (ROM), patient satisfaction, and improvement over time on patient reported outcome measures. This study will provide important information about the validity and reliability of using diaries to measure adherence to orthoses, and will be the first to provide objective data regarding the actual use of these orthoses and whether they help to decrease elbow stiffness.

DETAILED DESCRIPTION:
The elbow is prone to stiffness following trauma. Orthoses or splints are commonly used to manage this stiffness and prevent flexion contractures following elbow injury. One of the main orthoses used to treat patients who cannot extend their elbow following injury is to make an orthosis or splint to hold the elbow as straight as possible through the night to provide a gentle stretch. As patients gain the ability to straighten their elbow, the orthosis is reshaped over several weeks to continue to provide a stretch at night. This study will investigate the effectiveness of these orthoses for improving ROM, by correlating actual wearing time to ROM measurements. To date, there is no objective way of measuring whether patients actually wear these orthoses at night. Measurement of actual wearing time in the splint has been dependent on self-reported diaries to document wearing time.

The purpose of this study is to validate whether the use of a self-reported diary for orthosis use is accurate and valid. We will insert a temperature gauge into the orthosis during fabrication that measures temperature to an accuracy of one degree Celcius. This sensor is about the size of a watch battery, and patients will be told that it is measuring the force of stretch applied to the elbow, while in fact, it is measuring the amount of time that the orthosis is being worn. The temperature of the skin while wearing the orthosis heats up the sensor, and we can accurately predict (within 5 minutes of accuracy) how long the orthosis is worn each day.

We will have patients also fill out a self-report diary outlining how long they are wearing the orthosis each day, and compare these times to the measurements taken by the sensor. As a secondary outcome, we will look at whether the slightly different way the orthosis is made changes elbow stiffness via range of motion measurements of the elbow. Other data collected will include patient reported outcome measures including the Patient Rated Elbow Evaluation, The Disabilities of Arm, Shoulder, and Hand Questionnaire, and a patient satisfaction survey. This study will provide important information about the validity and reliability of using diaries to measure adherence to orthoses, and will be the first to provide objective data regarding the actual use of these orthoses and wearing time to changes in range of motion.

The Sensors are able to record 2 weeks on continuous data, and patients will be followed for 3 total visits - one for splint fabrication, at 2 weeks, 4 weeks, and 6 weeks, post splint fabrication. Patients will also attend regular therapy visits as needed, independent of these followups.

ELIGIBILITY:
Inclusion Criteria:

* All patients over age 18, with elbow trauma, referred by the Upper Limb Surgeons at the Roth McFarlane Hand & Upper Limb Centre (HULC) for night time extension splinting of the elbow following trauma

Exclusion Criteria:

* Elbow instability, infection, or other condition precluding the use of an extension orthosis at night time. Inability to wear the orthosis due to know skin reactions, claustrophobia, or ability to understand instructions and precautions provided in English. Patients will also be excluded if they are unable to return to HULC for follow up due to driving distance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over age 18, with elbow trauma, referred by the Upper Limb Surgeons at the Roth McFarlane Hand & Upper Limb Centre for night time extension splinting of the elbow following trauma. We will enroll patients consecutively.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Orthosis wearing time (sensor measured) | 6 weeks
  overall time in orthosis as measured by the sensor
Orthosis wearing time (self-reported) | 6 weeks
  overall time in orthosis reported by the patient

SECONDARY OUTCOMES:
Elbow ROM | 6 months
  goniometric measurement
Patient Rated Elbow Evaluation | 6 months
  patient reported outcome measure

IPD SHARING:
Plan to Share IPD: No